CLINICAL TRIAL: NCT02026934
Title: CliniMACS® CD34+ Reagent System for Expanded Access Use
Status: No longer available | Type: Expanded Access
Sponsor: Joseph Antin (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor-Investigator, Joseph Antin, Sponsor/Co-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Other Study IDs: 13-024
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Graft-Versus-Host Disease(GVHD); Anemia Due to Disturbance of Proliferation and/or Differentiation of Hematopoietic Stem Cells; Graft Failure; Delayed Graft Function
Keywords: Graft-Versus-Host Disease(GVHD); Hematopoietic Stem Cell Transplantation.; Graft failure; Graft exhaustion
MeSH Terms: conditions — Graft vs Host Disease; Delayed Graft Function

INTERVENTIONS:
Device: CliniMACS CD34 Reagent System — Following screening and enrollment, peripheral blood or bone marrow collection will be performed on the donor followed by subsequent CD34+ cell selection using the Miltenyi CliniMACS device. There is no limit to the number of CD34+ progenitors that can be administered. The CD34+ selected cells will be infused within 12 hours of the initiation of processing.

SUMMARY:
CliniMACs is an investigational device used to select and enrich stem cells. The device will select the stem cells with CD34+ protein. The participant will be infused with the CD34+ selected cells in the hopes that it will help the participant engraft. Engraftment is when transplanted stem cells resume production of healthy blood cells.

DETAILED DESCRIPTION:
* After the screening procedures confirm that the participant is eligible to participate in the research study: If the participant takes part in this research study, the participant (and their donor) will have the following tests and procedures:
* Donor Graft Collection: The participant's cell donor will undergo stem cell collection. The cells collected will be sent to the laboratory for processing.
* Donor Graft Processing: In the laboratory the CliniMACS device will be used to separate the CD34+ stem cells from the other types of cells in the graft. After completing the necessary safety tests, the CD34+ selected donor graft will be ready for administration.
* Donor Graft Infusion: The CD34+ selected donor graft will be infused through an intravenous (I.V.) catheter. The day of this infusion is called Day 0.
* Follow-Up Visits: Approximately 3, 6 and 12 months after the donor graft infusion, the participant will return to clinic for follow-up visits. At each of the visits, the participant will have a physical exam and asked questions about your general health. The participant will also have routine blood tests performed (approximately 1 tablespoon of blood).
* At times more cells are collected from a donation than are needed to do the transplantation. If your physician determines that it is preferable to administer a dose of cells that is less than the complete collection, the extra cells may be frozen and stored in our freezers for the participant's future use. If the cell counts do not improve, the participant will be given the remaining cells through an intravenous (I.V.) catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Diagnosis is graft exhaustion.
* Ability to understand and willingness to sign a written informed consent document
* Matched related or unrelated donor must consent to provide an allograft.

Exclusion Criteria:

* Symptomatic or uncontrolled cardiac failure or coronary artery disease.
* Karnofsky performance status < 60%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-03

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nikiforow, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States